CLINICAL TRIAL: NCT05877131
Title: Randomized Clinical Trial to Evaluate the Efficacy of Levobupivacaine 0.125% vs Ropivacaine 0.2%, in Hemodynamic Alterations in Pregnant Women in Labor and Their Fetal Repercussions
Brief Title: Evaluate Efficacy Levobupivacaine 0.125% Versuss Ropivacaine 0.2% in Hemodynamic Alterations in Labor and Fetal Repercussions
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Responsible Party: Principal Investigator, Mauricio Roberto Argañaraz Quinteros, Physician, Althaia Xarxa Assistencial Universitària de Manresa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEI-pendiente
Record Dates: First submitted 2023-03-20; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Hemodynamic Instability; Epidural; Pregnancy; Fetal Cardiac Disorder
Keywords: Hemodynamic instability; Epidural; Pregnancy; Fetal Cardiac disorder
MeSH Terms: interventions — Levobupivacaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levobupivacaina (Active Comparator): Levobupivacaine 0.125% , dosage 10 ml frequency 1 one dosis duration 1 hour
  Interventions: Drug: Levobupivacaine
- Ropivacaina (Active Comparator): Ropivacaine 2 % , dosage 10 ml frequency 1 one dosis duration 1 hour
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Levobupivacaine — To evaluate the efficacy of low-dose levobupivacaine (0.125%) (0.2) in avoiding hemodynamic changes after performing regional analgesia in pregnant women in labor and preventing changes in fetal heart rate and cardiotocographic recording.
  Arms: Levobupivacaina
Drug: Ropivacaine — To evaluate the efficacy of low-dose ropivacaine (0.2) in avoiding hemodynamic changes after performing regional analgesia in pregnant women in labor and preventing changes in fetal heart rate and cardiotocographic recording.
  Arms: Ropivacaina

SUMMARY:
INTRODUCTION:

Most studies on analgesia in pregnant women in labor mainly evaluate the effect of anesthetics on pain, mentioning hypotension as a side effect without investigating its impact on fetal well-being. The objective of the present study is to evaluate the efficacy of the use of low doses of local anesthetic (LA) to prevent hemodynamic alterations that manifest as a loss of fetal well-being.

METHODOLOGY/DESIGN:

It is a randomized clinical trial. Patients will be pregnant women in labor (dilation period) who want epidural anesthesia (EA), who will randomly receive 0.125% levobupivacaine (Group L) versus 0.2% ropivacaine (Group R). In both groups, controls of hemodynamic parameters and their relationship with changes in fetal heart rate (FHR) and cardiotocographic recording (RCTG) will be carried out during the first 60 minutes after the administration of the local anesthetic via the epidural route. In case of hypotension and/or subsequent FHR and RCTG alterations, they will also be recorded. The follow-up period will extend from the moment the patient enters the delivery room and requests epidural anesthesia until the moment the patient is discharged from the delivery room. The percentage of patients with hemodynamic alterations will be evaluated as a primary result, as well as the percentage of patients whose hemodynamic alterations are related to changes in FHR and RCTG, when using low doses of LA. In the following will also be evaluated in relation to analgesia, the onset time, level reached and degree of satisfaction; and various intra and postpartum side effects.

DISCUSSION:

Both groups of pregnant women in labor will be studied in order to obtain data on the potential impact of the use of low doses of local anesthetic via the epidural route on hemodynamic parameters and the state of well-being of the fetus.

DETAILED DESCRIPTION:
Any patient presenting in the delivery room or gynecology-obstetrics office of the hospital with prodromes, midwives or gynecologists will inform the principal investigator (PI). The IP will contact the patient to inform them of what the study consists of and if they wish to participate in it. In case of acceptance, the explanatory documentation and a questionnaire will be delivered to determine if it meets the inclusion criteria. If the pregnant patient at term meets the inclusion criteria, she is recruited to enter the study, it will also be used to resolve any doubts that the patient may have. Once the patient has signed the informed consent, the collaborating researcher (CI) of the recruiting center will be notified to contact the Althaia Innovation and Research Unit to find out the patient's assignment group. The collaborating researcher will be in charge of notifying the patient of the group to which she has been assigned (Intervention Group A or B).

Initially, the basal hemodynamic constants will be recorded: systolic blood pressure (SBP), mean blood pressure (TAM), diastolic blood pressure (TAD), pulse pressure (PP), systemic vascular resistance (SVR), cardiac output (CO), index Pulse Pressure Variation (PPV), Stroke Volume Variation (SVV), Heart Rate (HR), Stroke Volume (SV), Partial Pressure Oxygen Saturation (SpO2) via Clearsight device ®; pain score (VAS); degree of anxiety/depression by filling in a questionnaire to complete yourself; the degree of dilation. The FHR will also be recorded, as well as the different pathological patterns of the RCTG that appear, the Philips Avalon FM 30 monitor will be used for this.

The steps to follow for the administration of local anesthetic through the epidural catheter will be the following:

The mother's data (before and after AE) will be collected, including hemodynamic data: systolic blood pressure (SBP), mean blood pressure (TAM), diastolic blood pressure (TAD), pulse pressure (PP), vascular resistance heart rate (SVR), cardiac output (CO), cardiac index (CI), pulse pressure variation (PPV), stroke volume variation (VSV), heart rate (HR), stroke volume (SV), blood saturation partial pressure of oxygen (SpO2); pain score (VAS), degree of analgesia achieved, satisfaction obtained, time onset of analgesia, level of sensory block using the pin-prick test and the hot-cold test; degree of anxiety/depression by filling in a questionnaire to complete yourself; the degree of dilation. The fetal data (before and after the AE) of the FHR (values above or below the normal limits) will also be included, as well as the different pathological patterns of the RCTG that appear, due to hypotension or alterations. associated hemodynamics.

All pregnant women who will participate in this study will carry an intravenous cannula and will receive a fluid load of 500 cc. The position of the patients will be in a sitting position and the epidural puncture will be performed at the level of the L2-3 or L3-4 intervertebral space using a Tuohy 18 epidural needle. The loss of resistance technique with air or saline will be used according to the standards of our service.

A volume of 2 ml of 2% lidocaine will be administered via the epidural via the epidural catheter, after 3 minutes (it will be evaluated if undesirable effects appear: such as motor block due to accidental dural puncture, hypotension, nausea, vomiting), it will be administered to pregnant women the final volume (10 cc) of the local anesthetic randomly assigned via epidural.

After the administration of the initial bolus (Group A - Group B), the different constants or parameters to be evaluated will be recorded.

The measurement of the different hemodynamic variables will be recorded through a non-invasive device, the Clearsight®. The device will automatically determine the constants, which will be recorded at 5, 10, 15, 30, 45 and 60 minutes.

In the event of recording an episode of hypotension after the first 60 minutes, a record of all the hemodynamic variables evaluated will be made every 5 minutes for the following 60 minutes.

It will be determined which of the local anesthetics at low concentrations administered via the epidural is related to alteration of the hemodynamic parameters. To measure the different parameters, a non-invasive device (Clearsight) will be used, which will determine the existing hemodynamic alterations before, after, and during the first hour after the administration of the initial dose through the lumbar epidural catheter, as well as in the event of an episode. of hypotension or changes in FHR and/or RCTG after the first hour of catheter placement.

ELIGIBILITY:
Inclusion Criteria:

* - Woman > 18 years
* Request epidural anesthesia (EA)
* Expansion period
* Low obstetric risk
* ASA I-II (only one associated comorbidity, example: arterial hypertension, etc.)
* Cervix dilation ≥ 3
* single fetus
* Gestational age > 36 weeks
* Normal Fetal Heart Rate (110 -160 beats / minute)
* Normal Cardiotocographic record or absence of fetal heart rate patterns suggestive of risk of loss of fetal well-being or non-reassuring cardiotocographic record.

Exclusion Criteria:

* VAS ≤ 2
* Breech presentation
* Maternal fever > 38 years
* Pre-eclampsia and severe eclampsia
* Prenatal bleeding
* ASA II (more than one comorbidity)
* Chronic pain
* Substance abuse
* Contraindications for epidural analgesia (EA)
* Allergy to local anesthetics
* BMI >40 kg/m²
* Presence of RCTG not reassuring

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Systemic vascular resistance ( units of measure:dyn*s/cm5) | 10 minutes before epidural
  Systemic vascular resistance (SVR) is expressed by the equation: SVR = (MAP - CVP)/CO, where MAP is mean arterial pressure and CVP is central venous pressure.
Systemic vascular resistance ( units of measure:dyn*s/cm5) | 5 minutes after epidural
  Systemic vascular resistance (SVR) is expressed by the equation: SVR = (MAP - CVP)/CO, where MAP is mean arterial pressure and CVP is central venous pressure.
Systemic vascular resistance ( units of measure:dyn*s/cm5) | 10 minutes after epidural
  Systemic vascular resistance (SVR) is expressed by the equation: SVR = (MAP - CVP)/CO, where MAP is mean arterial pressure and CVP is central venous pressure.
Systemic vascular resistance ( units of measure:dyn*s/cm5) | 15 minutes after epidural
  Systemic vascular resistance (SVR) is expressed by the equation: SVR = (MAP - CVP)/CO, where MAP is mean arterial pressure and CVP is central venous pressure.
Systemic vascular resistance ( units of measure:dyn*s/cm5) | 30 minutes after epidural
  Systemic vascular resistance (SVR) is expressed by the equation: SVR = (MAP - CVP)/CO, where MAP is mean arterial pressure and CVP is central venous pressure.
Systemic vascular resistance ( units of measure:dyn*s/cm5) | 45 minutes after epidural
  Systemic vascular resistance (SVR) is expressed by the equation: SVR = (MAP - CVP)/CO, where MAP is mean arterial pressure and CVP is central venous pressure.
Systemic vascular resistance ( units of measure :dyn*s/cm5) | 60 minutes after epidural
  Systemic vascular resistance (SVR) is expressed by the equation: SVR = (MAP - CVP)/CO, where MAP is mean arterial pressure and CVP is central venous pressure.

SECONDARY OUTCOMES:
Systolic Blood Pressure (units of measure :mmHg) | 10 minutes before epidural
  Systolic pressure refers to the pressure of blood in the artery when the heart contracts. It is the upper (and highest) number in a blood pressure measurement.
Systolic Blood Pressure (units of measure :mmHg) | 5 minutes after epidural
  Systolic pressure refers to the pressure of blood in the artery when the heart contracts. It is the upper (and highest) number in a blood pressure measurement.
Systolic Blood Pressure (units of measure :mmHg) | 10 minutes after epidural
  Systolic pressure refers to the pressure of blood in the artery when the heart contracts. It is the upper (and highest) number in a blood pressure measurement.
Systolic Blood Pressure (units of measure :mmHg) | 15 minutes after epidural
  Systolic pressure refers to the pressure of blood in the artery when the heart contracts. It is the upper (and highest) number in a blood pressure measurement.
Systolic Blood Pressure (units of measure :mmHg) | 30 minutes after epidural
  Systolic pressure refers to the pressure of blood in the artery when the heart contracts. It is the upper (and highest) number in a blood pressure measurement.
Systolic Blood Pressure (units of measure :mmHg) | 45 minutes after epidural
  Systolic pressure refers to the pressure of blood in the artery when the heart contracts. It is the upper (and highest) number in a blood pressure measurement.
Systolic Blood Pressure (units of measure :mmHg) | 60 minutes after epidural
  Systolic pressure refers to the pressure of blood in the artery when the heart contracts. It is the upper (and highest) number in a blood pressure measurement.
Diastolic Blood Pressure (units of measure :mmHg) | 10 minutes before epidural
  Diastolic blood pressure refers to the pressure of blood in the artery when the heart relaxes between beats. It is the lower (and lower) number in a blood pressure measurement.
Diastolic Blood Pressure (units of measure :mmHg) | 5 minutes after epidural
  Diastolic blood pressure refers to the pressure of blood in the artery when the heart relaxes between beats. It is the lower (and lower) number in a blood pressure measurement.
Diastolic Blood Pressure (units of measure :mmHg) | 10 minutes after epidural
  Diastolic blood pressure refers to the pressure of blood in the artery when the heart relaxes between beats. It is the lower (and lower) number in a blood pressure measurement.
Diastolic Blood Pressure (units of measure :mmHg) | 15 minutes after epidural
  Diastolic blood pressure refers to the pressure of blood in the artery when the heart relaxes between beats. It is the lower (and lower) number in a blood pressure measurement.
Diastolic Blood Pressure (units of measure :mmHg) | 30 minutes after epidural
  Diastolic blood pressure refers to the pressure of blood in the artery when the heart relaxes between beats. It is the lower (and lower) number in a blood pressure measurement.
Diastolic Blood Pressure (units of measure :mmHg) | 45 minutes after epidural
  Diastolic blood pressure refers to the pressure of blood in the artery when the heart relaxes between beats. It is the lower (and lower) number in a blood pressure measurement.
Diastolic Blood Pressure (units of measure :mmHg) | 60 minutes after epidural
  Diastolic blood pressure refers to the pressure of blood in the artery when the heart relaxes between beats. It is the lower (and lower) number in a blood pressure measurement.
Mean Arterial Pressure (units of measure :mmHg) | 10 minutes before epidural
  Mean arterial pressure (MAP) is determined by cardiac output (CO), peripheral vascular resistance (PVR), and central venous pressure (CVP). The formula that integrates these concepts is:
  PAM = (GC x RVP) + PVC
Mean Arterial Pressure (units of measure :mmHg) | 5 minutes after epidural
  Mean arterial pressure (MAP) is determined by cardiac output (CO), peripheral vascular resistance (PVR), and central venous pressure (CVP). The formula that integrates these concepts is:
  PAM = (GC x RVP) + PVC
Mean Arterial Pressure (units of measure :mmHg) | 10 minutes after epidural
  Mean arterial pressure (MAP) is determined by cardiac output (CO), peripheral vascular resistance (PVR), and central venous pressure (CVP). The formula that integrates these concepts is:
  PAM = (GC x RVP) + PVC
Mean Arterial Pressure (units of measure :mmHg) | 15 minutes after epidural
  Mean arterial pressure (MAP) is determined by cardiac output (CO), peripheral vascular resistance (PVR), and central venous pressure (CVP). The formula that integrates these concepts is:
  PAM = (GC x RVP) + PVC
Mean Arterial Pressure (units of measure :mmHg) | 30 minutes after epidural
  Mean arterial pressure (MAP) is determined by cardiac output (CO), peripheral vascular resistance (PVR), and central venous pressure (CVP). The formula that integrates these concepts is:
  PAM = (GC x RVP) + PVC
Mean Arterial Pressure (units of measure :mmHg) | 45 minutes after epidural
  Mean arterial pressure (MAP) is determined by cardiac output (CO), peripheral vascular resistance (PVR), and central venous pressure (CVP). The formula that integrates these concepts is:
  PAM = (GC x RVP) + PVC
Mean Arterial Pressure (units of measure :mmHg) | 60 minutes after epidural
  Mean arterial pressure (MAP) is determined by cardiac output (CO), peripheral vascular resistance (PVR), and central venous pressure (CVP). The formula that integrates these concepts is:
  PAM = (GC x RVP) + PVC
Pulse Pressure (units of measure :mmHg) | 10 minutes before epidural
  Pulse pressure is the difference between systolic blood pressure (SBP) and diastolic blood pressure (DBP), and is an index of arterial compliance.
Pulse Pressure (units of measure :mmHg) | 5 minutes after epidural
  Pulse pressure is the difference between systolic blood pressure (SBP) and diastolic blood pressure (DBP), and is an index of arterial compliance.
Pulse Pressure (units of measure :mmHg) | 10 minutes after epidural
  Pulse pressure is the difference between systolic blood pressure (SBP) and diastolic blood pressure (DBP), and is an index of arterial compliance.
Pulse Pressure (units of measure :mmHg) | 15 minutes after epidural
  Pulse pressure is the difference between systolic blood pressure (SBP) and diastolic blood pressure (DBP), and is an index of arterial compliance.
Pulse Pressure (units of measure :mmHg) | 30 minutes after epidural
  Pulse pressure is the difference between systolic blood pressure (SBP) and diastolic blood pressure (DBP), and is an index of arterial compliance.
Pulse Pressure (units of measure :mmHg) | 45 minutes after epidural
  Pulse pressure is the difference between systolic blood pressure (SBP) and diastolic blood pressure (DBP), and is an index of arterial compliance.
Pulse Pressure (units of measure :mmHg) | 60 minutes after epidural
  Pulse pressure is the difference between systolic blood pressure (SBP) and diastolic blood pressure (DBP), and is an index of arterial compliance.
Cardiac Output (units of measure :L/min) | 10 minutes before epidural
  The volume of blood pumped from a ventricle each minute is known as cardiac output. It is the product of heart rate and stroke volume:
  Cardiac output = heart rate x stroke volume
Cardiac Output (units of measure :L/min) | 5 minutes after epidural
  The volume of blood pumped from a ventricle each minute is known as cardiac output. It is the product of heart rate and stroke volume:
  Cardiac output = heart rate x stroke volume
Cardiac Output (units of measure :L/min) | 10 minutes after epidural
  The volume of blood pumped from a ventricle each minute is known as cardiac output. It is the product of heart rate and stroke volume:
  Cardiac output = heart rate x stroke volume
Cardiac Output (units of measure :L/min) | 15 minutes after epidural
  The volume of blood pumped from a ventricle each minute is known as cardiac output. It is the product of heart rate and stroke volume:
  Cardiac output = heart rate x stroke volume
Cardiac Output (units of measure :L/min) | 30 minutes after epidural
  The volume of blood pumped from a ventricle each minute is known as cardiac output. It is the product of heart rate and stroke volume:
  Cardiac output = heart rate x stroke volume
Cardiac Output (units of measure :L/min) | 45 minutes after epidural
  The volume of blood pumped from a ventricle each minute is known as cardiac output. It is the product of heart rate and stroke volume:
  Cardiac output = heart rate x stroke volume
Cardiac Output (units of measure :L/min) | 60 minutes after epidural
  The volume of blood pumped from a ventricle each minute is known as cardiac output. It is the product of heart rate and stroke volume:
  Cardiac output = heart rate x stroke volume
Cardiac Index ( units of measure :L/min/m2) | 10 minutes before epidural
  A cardio dynamic measure based on the cardiac output, which is the amount of blood the left ventricle ejects into the systemic circulation in one minute, measured in liters per minute (l/min). Cardiac output is indexed to a patient's body size by dividing by the body surface area to yield the cardiac index.
  Cardiac Index = Cardiac Output / Body Surface Area = (Heart Rate * Stroke Volume) / Body Surface Area
Cardiac Index ( units of measure :L/min/m2) | 5 minutes after epidural
  A cardio dynamic measure based on the cardiac output, which is the amount of blood the left ventricle ejects into the systemic circulation in one minute, measured in liters per minute (l/min). Cardiac output is indexed to a patient's body size by dividing by the body surface area to yield the cardiac index.
  Cardiac Index = Cardiac Output / Body Surface Area = (Heart Rate * Stroke Volume) / Body Surface Area
Cardiac Index ( units of measure :L/min/m2) | 10 minutes after epidural
  A cardio dynamic measure based on the cardiac output, which is the amount of blood the left ventricle ejects into the systemic circulation in one minute, measured in liters per minute (l/min). Cardiac output is indexed to a patient's body size by dividing by the body surface area to yield the cardiac index.
  Cardiac Index = Cardiac Output / Body Surface Area = (Heart Rate * Stroke Volume) / Body Surface Area
Cardiac Index ( units of measure :L/min/m2) | 15 minutes after epidural
  A cardio dynamic measure based on the cardiac output, which is the amount of blood the left ventricle ejects into the systemic circulation in one minute, measured in liters per minute (l/min). Cardiac output is indexed to a patient's body size by dividing by the body surface area to yield the cardiac index.
  Cardiac Index = Cardiac Output / Body Surface Area = (Heart Rate * Stroke Volume) / Body Surface Arealimits) will also be included
Cardiac Index ( units of measure :L/min/m2) | 30 minutes after epidural
  A cardio dynamic measure based on the cardiac output, which is the amount of blood the left ventricle ejects into the systemic circulation in one minute, measured in liters per minute (l/min). Cardiac output is indexed to a patient's body size by dividing by the body surface area to yield the cardiac index.
  Cardiac Index = Cardiac Output / Body Surface Area = (Heart Rate * Stroke Volume) / Body Surface Area
Cardiac Index ( units of measure :L/min/m2) | 45 minutes after epidural
  A cardio dynamic measure based on the cardiac output, which is the amount of blood the left ventricle ejects into the systemic circulation in one minute, measured in liters per minute (l/min). Cardiac output is indexed to a patient's body size by dividing by the body surface area to yield the cardiac index.
  Cardiac Index = Cardiac Output / Body Surface Area = (Heart Rate * Stroke Volume) / Body Surface Area
Cardiac Index ( units of measure :L/min/m2) | 60 minutes after epidural
  A cardio dynamic measure based on the cardiac output, which is the amount of blood the left ventricle ejects into the systemic circulation in one minute, measured in liters per minute (l/min). Cardiac output is indexed to a patient's body size by dividing by the body surface area to yield the cardiac index.
  Cardiac Index = Cardiac Output / Body Surface Area = (Heart Rate * Stroke Volume) / Body Surface Area
Pulse Pressure Variation ( units of measure :% Percent) | 10 minutes before epidural
  Pulse pressure variation (PPV) is an effective and widely used dynamic parameter to predict the increase in cardiac output after fluid administration. Ideally, PPV measurement should be performed with a closed chest and mechanical ventilation with a tidal volume of 8 mL/kg.PPV was calculated as the percentage changes in arterial pulse pressure during a ventilatory cycle as [(PPmax - PPmin)/(PPmax
  + PPmin)/2] × 100, where PPmax and PPmin represent the maximal and minimal arterial pulse pressure, respectively
Pulse Pressure Variation ( units of measure :% Percent) | 5 minutes after epidural
  Pulse pressure variation (PPV) is an effective and widely used dynamic parameter to predict the increase in cardiac output after fluid administration. Ideally, PPV measurement should be performed with a closed chest and mechanical ventilation with a tidal volume of 8 mL/kg.PPV was calculated as the percentage changes in arterial pulse pressure during a ventilatory cycle as [(PPmax - PPmin)/(PPmax
  + PPmin)/2] × 100, where PPmax and PPmin represent the maximal and minimal arterial pulse pressure, respectively
Pulse Pressure Variation ( units of measure :% Percent) | 10 minutes after epidural
  Pulse pressure variation (PPV) is an effective and widely used dynamic parameter to predict the increase in cardiac output after fluid administration. Ideally, PPV measurement should be performed with a closed chest and mechanical ventilation with a tidal volume of 8 mL/kg.PPV was calculated as the percentage changes in arterial pulse pressure during a ventilatory cycle as [(PPmax - PPmin)/(PPmax
  + PPmin)/2] × 100, where PPmax and PPmin represent the maximal and minimal arterial pulse pressure, respectively
Pulse Pressure Variation ( units of measure :% Percent) | 15 minutes after epidural
  Pulse pressure variation (PPV) is an effective and widely used dynamic parameter to predict the increase in cardiac output after fluid administration. Ideally, PPV measurement should be performed with a closed chest and mechanical ventilation with a tidal volume of 8 mL/kg.PPV was calculated as the percentage changes in arterial pulse pressure during a ventilatory cycle as [(PPmax - PPmin)/(PPmax
  + PPmin)/2] × 100, where PPmax and PPmin represent the maximal and minimal arterial pulse pressure, respectively
Pulse Pressure Variation ( units of measure :% Percent) | 30 minutes after epidural
  Pulse pressure variation (PPV) is an effective and widely used dynamic parameter to predict the increase in cardiac output after fluid administration. Ideally, PPV measurement should be performed with a closed chest and mechanical ventilation with a tidal volume of 8 mL/kg.PPV was calculated as the percentage changes in arterial pulse pressure during a ventilatory cycle as [(PPmax - PPmin)/(PPmax
  + PPmin)/2] × 100, where PPmax and PPmin represent the maximal and minimal arterial pulse pressure, respectively
Pulse Pressure Variation ( units of measure :% Percent) | 45 minutes after epidural
  Pulse pressure variation (PPV) is an effective and widely used dynamic parameter to predict the increase in cardiac output after fluid administration. Ideally, PPV measurement should be performed with a closed chest and mechanical ventilation with a tidal volume of 8 mL/kg.PPV was calculated as the percentage changes in arterial pulse pressure during a ventilatory cycle as [(PPmax - PPmin)/(PPmax
  + PPmin)/2] × 100, where PPmax and PPmin represent the maximal and minimal arterial pulse pressure, respectively
Pulse Pressure Variation ( units of measure :% Percent) | 60 minutes after epidural
  Pulse pressure variation (PPV) is an effective and widely used dynamic parameter to predict the increase in cardiac output after fluid administration. Ideally, PPV measurement should be performed with a closed chest and mechanical ventilation with a tidal volume of 8 mL/kg.PPV was calculated as the percentage changes in arterial pulse pressure during a ventilatory cycle as [(PPmax - PPmin)/(PPmax
  + PPmin)/2] × 100, where PPmax and PPmin represent the maximal and minimal arterial pulse pressure, respectively
(Maternal) Heart Rate (units of measure: beats per minute) | 10 minutes before epidural
  The number of times the heart beats during a certain period, usually one minute.
  The resting heart rate normally ranges from 60 to 100 beats per minute in a healthy adult at rest.
(Maternal) Heart Rate (units of measure: beats per minute) | 5 minutes after epidural
  The number of times the heart beats during a certain period, usually one minute.
  The resting heart rate normally ranges from 60 to 100 beats per minute in a healthy adult at rest.
(Maternal) Heart Rate (units of measure: beats per minute) | 10 minutes after epidural
  The number of times the heart beats during a certain period, usually one minute.
  The resting heart rate normally ranges from 60 to 100 beats per minute in a healthy adult at rest.
(Maternal) Heart Rate (units of measure: beats per minute) | 15 minutes after epidural
  The number of times the heart beats during a certain period, usually one minute.
  The resting heart rate normally ranges from 60 to 100 beats per minute in a healthy adult at rest.
(Maternal) Heart Rate (units of measure: beats per minute) | 30 minutes after epidural
  The number of times the heart beats during a certain period, usually one minute.
  The resting heart rate normally ranges from 60 to 100 beats per minute in a healthy adult at rest.
(Maternal) Heart Rate (units of measure: beats per minute) | 45 minutes after epidural
  The number of times the heart beats during a certain period, usually one minute.
  The resting heart rate normally ranges from 60 to 100 beats per minute in a healthy adult at rest.
(Maternal) Heart Rate (units of measure: beats per minute) | 60 minutes after epidural
  The number of times the heart beats during a certain period, usually one minute.
  The resting heart rate normally ranges from 60 to 100 beats per minute in a healthy adult at rest.
Stroke Volume (units of measure :ml) | 10 minutes before epidural
  Stroke volume is the volume of blood pumped out of the left ventricle of the heart during each systolic cardiac contraction. The SV volume may be calculated as the difference between the left ventricular end-diastolic volume and the left ventricular end-systolic volume (ESV).
Stroke Volume (units of measure :ml) | 5 minutes after epidural
  Stroke volume is the volume of blood pumped out of the left ventricle of the heart during each systolic cardiac contraction. The SV volume may be calculated as the difference between the left ventricular end-diastolic volume and the left ventricular end-systolic volume (ESV).
Stroke Volume (units of measure :ml) | 10 minutes after epidural
  Stroke volume is the volume of blood pumped out of the left ventricle of the heart during each systolic cardiac contraction. The SV volume may be calculated as the difference between the left ventricular end-diastolic volume and the left ventricular end-systolic volume (ESV).
Stroke Volume (units of measure :ml) | 15 minutes after epidural
  Stroke volume is the volume of blood pumped out of the left ventricle of the heart during each systolic cardiac contraction. The SV volume may be calculated as the difference between the left ventricular end-diastolic volume and the left ventricular end-systolic volume (ESV).
Stroke Volume (units of measure :ml) | 30 minutes after epidural
  Stroke volume is the volume of blood pumped out of the left ventricle of the heart during each systolic cardiac contraction. The SV volume may be calculated as the difference between the left ventricular end-diastolic volume and the left ventricular end-systolic volume (ESV).
Stroke Volume (units of measure :ml) | 45 minutes after epidural
  Stroke volume is the volume of blood pumped out of the left ventricle of the heart during each systolic cardiac contraction. The SV volume may be calculated as the difference between the left ventricular end-diastolic volume and the left ventricular end-systolic volume (ESV).
Stroke Volume (units of measure :ml) | 60 minutes after epidural
  Stroke volume is the volume of blood pumped out of the left ventricle of the heart during each systolic cardiac contraction. The SV volume may be calculated as the difference between the left ventricular end-diastolic volume and the left ventricular end-systolic volume (ESV).
Systolic Variation Volume ( units of measure :% Percent) | 10 minutes before epidural
  Stroke volume variation (SVV) has been shown to be a reliable predictor of fluid responsiveness.SVV is assessed using the following equation: SVV (%) = (SVmax - SVmin)/SVmean
Systolic Variation Volume ( units of measure :% Percent) | 5 minutes after epidural
  Stroke volume variation (SVV) has been shown to be a reliable predictor of fluid responsiveness.SVV is assessed using the following equation: SVV (%) = (SVmax - SVmin)/SVmean
Systolic Variation Volume ( units of measure :% Percent) | 10 minutes after epidural
  Stroke volume variation (SVV) has been shown to be a reliable predictor of fluid responsiveness.SVV is assessed using the following equation: SVV (%) = (SVmax - SVmin)/SVmean
Systolic Variation Volume ( units of measure :% Percent) | 15 minutes after epidural
  Stroke volume variation (SVV) has been shown to be a reliable predictor of fluid responsiveness.SVV is assessed using the following equation: SVV (%) = (SVmax - SVmin)/SVmean
Systolic Variation Volume ( units of measure :% Percent) | 30 minutes after epidural
  Stroke volume variation (SVV) has been shown to be a reliable predictor of fluid responsiveness.SVV is assessed using the following equation: SVV (%) = (SVmax - SVmin)/SVmean
Systolic Variation Volume ( units of measure :% Percent) | 45 minutes after epidural
  Stroke volume variation (SVV) has been shown to be a reliable predictor of fluid responsiveness.SVV is assessed using the following equation: SVV (%) = (SVmax - SVmin)/SVmean
Systolic Variation Volume ( units of measure :% Percent) | 60 minutes after epidural
  Stroke volume variation (SVV) has been shown to be a reliable predictor of fluid responsiveness.SVV is assessed using the following equation: SVV (%) = (SVmax - SVmin)/SVmean
Arterial Oxigen Saturation ( units of measure :% Percent) | 10 minutes before epidural
  Arterial oxygen saturation (SaO2) is a measure of hemoglobin oxygenation in the arterial compartment of the circulatory system. It is not a measure of the total oxygen content in the arterial blood because a small fraction of oxygen (about 2%) is dissolved in the plasma. To determine overall oxygen-carrying capacity of the blood, multiply 1.34 ml/g by the patient's hemoglobin level in g/dL and by Spo2.
Arterial Oxigen Saturation ( units of measure :% Percent) | 5 minutes after epidural
  Arterial oxygen saturation (SaO2) is a measure of hemoglobin oxygenation in the arterial compartment of the circulatory system. It is not a measure of the total oxygen content in the arterial blood because a small fraction of oxygen (about 2%) is dissolved in the plasma. To determine overall oxygen-carrying capacity of the blood, multiply 1.34 ml/g by the patient's hemoglobin level in g/dL and by Spo2.
Arterial Oxigen Saturation ( units of measure :% Percent) | 10 minutes after epidural
  Arterial oxygen saturation (SaO2) is a measure of hemoglobin oxygenation in the arterial compartment of the circulatory system. It is not a measure of the total oxygen content in the arterial blood because a small fraction of oxygen (about 2%) is dissolved in the plasma. To determine overall oxygen-carrying capacity of the blood, multiply 1.34 ml/g by the patient's hemoglobin level in g/dL and by Spo2.
Arterial Oxigen Saturation ( units of measure :% Percent) | 15 minutes after epidural
  Arterial oxygen saturation (SaO2) is a measure of hemoglobin oxygenation in the arterial compartment of the circulatory system. It is not a measure of the total oxygen content in the arterial blood because a small fraction of oxygen (about 2%) is dissolved in the plasma. To determine overall oxygen-carrying capacity of the blood, multiply 1.34 ml/g by the patient's hemoglobin level in g/dL and by Spo2.
Arterial Oxigen Saturation ( units of measure :% Percent) | 30 minutes after epidural
  Arterial oxygen saturation (SaO2) is a measure of hemoglobin oxygenation in the arterial compartment of the circulatory system. It is not a measure of the total oxygen content in the arterial blood because a small fraction of oxygen (about 2%) is dissolved in the plasma. To determine overall oxygen-carrying capacity of the blood, multiply 1.34 ml/g by the patient's hemoglobin level in g/dL and by Spo2.
Arterial Oxigen Saturation ( units of measure :% Percent) | 45 minutes after epidural
  Arterial oxygen saturation (SaO2) is a measure of hemoglobin oxygenation in the arterial compartment of the circulatory system. It is not a measure of the total oxygen content in the arterial blood because a small fraction of oxygen (about 2%) is dissolved in the plasma. To determine overall oxygen-carrying capacity of the blood, multiply 1.34 ml/g by the patient's hemoglobin level in g/dL and by Spo2.
Arterial Oxigen Saturation ( units of measure :% Percent) | 60 minutes after epidural
  Arterial oxygen saturation (SaO2) is a measure of hemoglobin oxygenation in the arterial compartment of the circulatory system. It is not a measure of the total oxygen content in the arterial blood because a small fraction of oxygen (about 2%) is dissolved in the plasma. To determine overall oxygen-carrying capacity of the blood, multiply 1.34 ml/g by the patient's hemoglobin level in g/dL and by Spo2.
Fetal heart rate (units of measure: beats per minute) | 10 minutes before epidural
  The average fetal heart rate is between 110 and 160 beats per minute. It can vary by 5 to 25 beats per minute. The fetal heart rate may change by differents conditions in the uterus. An abnormal fetal heart rate may mean that is not getting enough oxygen or that there are other problems.
Fetal heart rate (units of measure: beats per minute) | 5 minutes after epidural
  The average fetal heart rate is between 110 and 160 beats per minute. It can vary by 5 to 25 beats per minute. The fetal heart rate may change by differents conditions in the uterus. An abnormal fetal heart rate may mean that is not getting enough oxygen or that there are other problems.
Fetal heart rate (units of measure: beats per minute) | 10 minutes after epidural
  The average fetal heart rate is between 110 and 160 beats per minute. It can vary by 5 to 25 beats per minute. The fetal heart rate may change by differents conditions in the uterus. An abnormal fetal heart rate may mean that is not getting enough oxygen or that there are other problems.
Fetal heart rate (units of measure: beats per minute) | 15 minutes after epidural
  The average fetal heart rate is between 110 and 160 beats per minute. It can vary by 5 to 25 beats per minute. The fetal heart rate may change by differents conditions in the uterus. An abnormal fetal heart rate may mean that is not getting enough oxygen or that there are other problems.
Fetal heart rate (units of measure: beats per minute) | 30 minutes after epidural
  The average fetal heart rate is between 110 and 160 beats per minute. It can vary by 5 to 25 beats per minute. The fetal heart rate may change by differents conditions in the uterus. An abnormal fetal heart rate may mean that is not getting enough oxygen or that there are other problems.
Fetal heart rate (units of measure: beats per minute) | 45 minutes after epidural
  The average fetal heart rate is between 110 and 160 beats per minute. It can vary by 5 to 25 beats per minute. The fetal heart rate may change by differents conditions in the uterus. An abnormal fetal heart rate may mean that is not getting enough oxygen or that there are other problems.
Fetal heart rate (units of measure: beats per minute) | 60 minutes after epidural
  The average fetal heart rate is between 110 and 160 beats per minute. It can vary by 5 to 25 beats per minute. The fetal heart rate may change by differents conditions in the uterus. An abnormal fetal heart rate may mean that is not getting enough oxygen or that there are other problems.
Variability (units of measure: beats per minute) | 10 minutes before epidural
  This the minor fluctuation in baseline FHR. It is assessed by estimating the difference in bpm between the highest peak and lowest trough of fluctuation in one minute segments of the trace
Variability (units of measure: beats per minute) | 5 minutes after epidural
  This the minor fluctuation in baseline FHR. It is assessed by estimating the difference in bpm between the highest peak and lowest trough of fluctuation in one minute segments of the trace
Variability (units of measure: beats per minute) | 10 minutes after epidural
  This the minor fluctuation in baseline FHR. It is assessed by estimating the difference in bpm between the highest peak and lowest trough of fluctuation in one minute segments of the trace
Variability (units of measure: beats per minute) | 15 minutes after epidural
  This the minor fluctuation in baseline FHR. It is assessed by estimating the difference in bpm between the highest peak and lowest trough of fluctuation in one minute segments of the trace
Variability (units of measure: beats per minute) | 30 minutes after epidural
  This the minor fluctuation in baseline FHR. It is assessed by estimating the difference in bpm between the highest peak and lowest trough of fluctuation in one minute segments of the trace
Variability (units of measure: beats per minute) | 45 minutes after epidural
  This the minor fluctuation in baseline FHR. It is assessed by estimating the difference in bpm between the highest peak and lowest trough of fluctuation in one minute segments of the trace
Variability (units of measure: beats per minute) | 60 minutes after epidural
  This the minor fluctuation in baseline FHR. It is assessed by estimating the difference in bpm between the highest peak and lowest trough of fluctuation in one minute segments of the trace
Accelerations (units of measure: beats per minute) | 10 minutes before epidural
  These are transient increases in FHR of 15bpm or more above the baseline and lasting 15 seconds.
Accelerations (units of measure: beats per minute) | 5 minutes after epidural
  These are transient increases in FHR of 15bpm or more above the baseline and lasting 15 seconds.
Accelerations (units of measure: beats per minute) | 10 minutes after epidural
  These are transient increases in FHR of 15bpm or more above the baseline and lasting 15 seconds.
Accelerations (units of measure: beats per minute) | 15 minutes after epidural
  These are transient increases in FHR of 15bpm or more above the baseline and lasting 15 seconds.
Accelerations (units of measure: beats per minute) | 30 minutes after epidural
  These are transient increases in FHR of 15bpm or more above the baseline and lasting 15 seconds.
Accelerations (units of measure: beats per minute) | 45 minutes after epidural
  These are transient increases in FHR of 15bpm or more above the baseline and lasting 15 seconds.
Accelerations (units of measure: beats per minute) | 60 minutes after epidural
  These are transient increases in FHR of 15bpm or more above the baseline and lasting 15 seconds.
Decelerations (units of measure: beats per minute) | 10 minutes before epidural
  These are transient episodes of decrease of FHR below the baseline of more than 15 bpm lasting at least 15 seconds.
Decelerations (units of measure: beats per minute) | 5 minutes after epidural
  These are transient episodes of decrease of FHR below the baseline of more than 15 bpm lasting at least 15 seconds.
Decelerations (units of measure: beats per minute) | 10 minutes after epidural
  These are transient episodes of decrease of FHR below the baseline of more than 15 bpm lasting at least 15 seconds.
Decelerations (units of measure: beats per minute) | 15 minutes after epidural
  These are transient episodes of decrease of FHR below the baseline of more than 15 bpm lasting at least 15 seconds.
Decelerations (units of measure: beats per minute) | 30 minutes after epidural
  These are transient episodes of decrease of FHR below the baseline of more than 15 bpm lasting at least 15 seconds.
Decelerations (units of measure: beats per minute) | 45 minutes after epidural
  These are transient episodes of decrease of FHR below the baseline of more than 15 bpm lasting at least 15 seconds.
Decelerations (units of measure: beats per minute) | 60 minutes after epidural
  These are transient episodes of decrease of FHR below the baseline of more than 15 bpm lasting at least 15 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Althaia Xarxa Assitensial i Universitaria Manresa, Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ACOG Committee on Practice Bulletins. ACOG practice bulletin. Clinical management guidelines for obstetrician-gynecologists. Number 44, July 2003. (Replaces Committee Opinion Number 252, March 2001). Obstet Gynecol. 2003 Jul;102(1):203-13. No abstract available. PMID 12850637
- [Background] Preston R, Crosby ET, Kotarba D, Dudas H, Elliott RD. Maternal positioning affects fetal heart rate changes after epidural analgesia for labour. Can J Anaesth. 1993 Dec;40(12):1136-41. doi: 10.1007/BF03009602. PMID 8281589
- [Background] Lappen JR, Chien EK, Mercer BM. Contraction-Associated Maternal Heart Rate Decelerations: A Pragmatic Marker of Intrapartum Volume Status. Obstet Gynecol. 2018 Oct;132(4):1011-1017. doi: 10.1097/AOG.0000000000002808. PMID 30130346
- [Background] Valensise H, Lo Presti D, Tiralongo GM, Pisani I, Gagliardi G, Vasapollo B, Frigo MG. Foetal heart rate deceleration with combined spinal-epidural analgesia during labour: a maternal haemodynamic cardiac study. J Matern Fetal Neonatal Med. 2016;29(12):1980-6. doi: 10.3109/14767058.2015.1072156. Epub 2015 Aug 28. PMID 26333691
- [Background] Collins KM, Bevan DR, Beard RW. Fluid loading to reduce abnormalities of fetal heart rate and maternal hypotension during epidural analgesia in labour. Br Med J. 1978 Nov 25;2(6150):1460-1. doi: 10.1136/bmj.2.6150.1460. PMID 719463
- [Background] Umstad MP, Ross A, Rushford DD, Permezel M. Epidural analgesia and fetal heart rate abnormalities. Aust N Z J Obstet Gynaecol. 1993 Aug;33(3):269-72. doi: 10.1111/j.1479-828x.1993.tb02083.x. PMID 8304890
- [Background] Kubli M, Shennan AH, Seed PT, O'Sullivan G. A randomised controlled trial of fluid pre-loading before low dose epidural analgesia for labour. Int J Obstet Anesth. 2003 Oct;12(4):256-60. doi: 10.1016/S0959-289X(03)00071-2. PMID 15321453
- [Background] Hofmeyr G, Cyna A, Middleton P. Prophylactic intravenous preloading for regional analgesia in labour. Cochrane Database Syst Rev. 2004 Oct 18;2004(4):CD000175. doi: 10.1002/14651858.CD000175.pub2. PMID 15494990
- [Background] Peyronnet V, Roses A, Girault A, Bonnet MP, Goffinet F, Tsatsaris V, Lecarpentier E. Lower limbs venous compression reduces the incidence of maternal hypotension following epidural analgesia during term labor. Eur J Obstet Gynecol Reprod Biol. 2017 Dec;219:94-99. doi: 10.1016/j.ejogrb.2017.10.016. Epub 2017 Oct 16. PMID 29073508